CLINICAL TRIAL: NCT04716166
Title: Compare the Effects of Volume-oriented Versus Flow-oriented Incentive Spirometry on Pulmonary Function and Functional Capacity in Patients of Upper Abdominal Laparoscopic Surgery
Brief Title: Incentive Spirometry and Upper Abdominal Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Muhammad Shakir Khan
Record Dates: First submitted 2021-01-19; First posted 2021-01-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Cholecystitis; Perforated Duodenal Ulcer; Diaphragmatic Hernia; Benign Pancreas Tumor; Malignant Pancreatic Neoplasm; Splenic Infarction; Splenomegaly; Choledocholithiasis; Hiatal Hernia
Keywords: Flow oriented incentive spirometry; Volume oriented incentive spirometry; Digital spirometer; Six minute walk test; Forced vital capacity (FVC); Forced Expiratory Volume in the first second (FEV1); Upper abdominal laparoscopy
MeSH Terms: conditions — Cholecystitis; Hernia, Diaphragmatic; Pancreatic Neoplasms; Splenic Infarction; Splenomegaly; Choledocholithiasis; Hernia, Hiatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volume-oriented incentive spirometry (Experimental): Postoperative Volume oriented incentive spirometry 3 times a day
  Interventions: Other: Volume-oriented incentive spirometry
- Flow-oriented incentive spirometry (Experimental): Postoperative Flow oriented incentive spirometry 3 times a day
  Interventions: Other: Flow-oriented incentive spirometry

INTERVENTIONS:
Other: Volume-oriented incentive spirometry — 3 sets of 5 repeated deep breaths using volume oriented incentive spirometry 3 times a day for 2 days
  Arms: Volume-oriented incentive spirometry
Other: Flow-oriented incentive spirometry — 3 sets of 5 repeated deep breaths using flow oriented incentive spirometry 3 times a day for 2 days
  Arms: Flow-oriented incentive spirometry

SUMMARY:
To compare the effects of volume-oriented versus flow-oriented incentive spirometry on pulmonary function tests and functional capacity in patients of upper abdominal laparoscopic surgery. Previous studies were designed to target only spirometer without focusing on its different types and their effects. This study covers the research gap and therefore is designed to observe effects of different types of spirometer on pulmonary function of patients undergoing upper abdominal laparoscopic surgery.

DETAILED DESCRIPTION:
The volume oriented incentive spirometer enables the patient to inhale air through a mouthpiece and corrugated tubing which is attached to a plastic bellows. The volume of air displaced is indicated on a scale located on the device enclosure. After the patient has achieved the maximum volume, the individual is instructed to hold this volume constant for 3 to 5 seconds.

Studies suggest a physiologically significant difference in the effect of the flow- and volume-oriented incentive spirometer. Flow-oriented devices enforce more work of breathing and increase muscular activity of the upper chest. Volume-oriented devices enforce less work of breathing and improve diaphragmatic activity.

Research was carried out a study on two experimental groups of patients in order to evaluate the effects of aerobic exercise training and incentive spirometry in controlling pulmonary complications following laparoscopic cholecystectomy, results indicated a significant reduction in heart rate, Oxygen Saturation of hemoglobin (SaO2), and inspiratory capacity for both groups. The researchers concluded that aerobic exercise and incentive spirometry were beneficial in reducing the postoperative pulmonary complications after laparoscopic cholecystectomy.

Another study observed the comparative study on the effect of preoperative and postoperative incentive spirometry on the pulmonary function of fifty patients who had undergone laparoscopic cholecystectomy. The authors concluded that pulmonary function is well-preserved with preoperative than postoperative incentive spirometry.

Another study observed that the volume incentive spirometry resulted in early recovery of both pulmonary function and diaphragm movement in patients who undergone laparoscopic abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient with upper abdominal surgery (laparoscopy)

Exclusion Criteria:

* Patients who had undergone open abdominal surgery and laparoscopic obstetrics and gynecological surgery.
* Patients with unstable hemodynamic parameters (arterial pressure<100 mmHg systolic and <60 mmHg for diastolic and mean arterial Pressure (MAP) <80mmHg.
* Patients with postoperative complications requiring mechanical ventilation.
* Uncooperative patients or patients unable to understand or to use the device properly
* Recent history of lower extremity fracture

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Functional Capacity | 2 days
  The six-minute walk test (6MWT) is a submaximal exercise test for evaluating physical functional capacity. Six meter walk distance ranges from 400 to 700 meter in normal individuals
Total Lung Capacity | 2 days
  Changes from the baseline will be measured on daily basis. Pulmonary function test will be measured by using a digital spirometer. Spirometry assesses the integrated mechanical function of the lung, chest wall, respiratory muscles, and airways by measuring the total volume of air exhaled from a full lung total lung capacity [TLC] TLC has a normal value ranges from 80% to 120%, of the predicted ratio.
Forced vital capacity (FVC) | 2 days
  Changes from the baseline will be measured on daily basis. Pulmonary function test will be measured by using a digital spirometer. FVC is the total volume of air that can be exhaled during a maximally forced expiration effort. It ranges from 80% to 120% of the predicted value.
Forced expiratory volume in 1 second (FEV1) | 2 days
  FEV1 is the volume of air that can forcibly be blown out in the first 1 second, after full inspiration. Average values for FEV1 in healthy people depend mainly on sex and age. Values of between 80% and 120% of the average value are considered normal.
FEV1/FVC ratio | 2 days
  FEEV1/FVC is the ratio of FEV1 to FVC. In healthy adults, this should be approximately 70-80%

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Fatima, MSPT-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Railway General hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alaparthi GK, Augustine AJ, Anand R, Mahale A. Comparison of Diaphragmatic Breathing Exercise, Volume and Flow Incentive Spirometry, on Diaphragm Excursion and Pulmonary Function in Patients Undergoing Laparoscopic Surgery: A Randomized Controlled Trial. Minim Invasive Surg. 2016;2016:1967532. doi: 10.1155/2016/1967532. Epub 2016 Jul 21. PMID 27525116
- [Background] do Nascimento Junior P, Modolo NS, Andrade S, Guimaraes MM, Braz LG, El Dib R. Incentive spirometry for prevention of postoperative pulmonary complications in upper abdominal surgery. Cochrane Database Syst Rev. 2014 Feb 8;2014(2):CD006058. doi: 10.1002/14651858.CD006058.pub3. PMID 24510642
- [Background] Kundra P, Vitheeswaran M, Nagappa M, Sistla S. Effect of preoperative and postoperative incentive spirometry on lung functions after laparoscopic cholecystectomy. Surg Laparosc Endosc Percutan Tech. 2010 Jun;20(3):170-2. doi: 10.1097/SLE.0b013e3181db81ce. PMID 20551816
- [Background] Soares SM, Jannuzzi HP, Kassab MF, Nucci LB, Paschoal MA. Investigation of the immediate pre-operative physical capacity of patients scheduled for elective abdominal surgery using the 6-minute walk test. Physiotherapy. 2015 Sep;101(3):292-7. doi: 10.1016/j.physio.2014.11.004. Epub 2014 Dec 17. PMID 25721252
- [Background] Kumar AS, Alaparthi GK, Augustine AJ, Pazhyaottayil ZC, Ramakrishna A, Krishnakumar SK. Comparison of Flow and Volume Incentive Spirometry on Pulmonary Function and Exercise Tolerance in Open Abdominal Surgery: A Randomized Clinical Trial. J Clin Diagn Res. 2016 Jan;10(1):KC01-6. doi: 10.7860/JCDR/2016/16164.7064. Epub 2016 Jan 1. PMID 26894090